CLINICAL TRIAL: NCT05179330
Title: Visual Feedback in Lower Limb Rehabilitation: the Alpha and the OMEGO®
Brief Title: Visual Feedback in Lower Limb Rehabilitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, PADUA LUCA, Associated Professor, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 3515
Record Dates: First submitted 2021-12-02; First posted 2022-01-05 (Actual); Last update posted 2024-02-22 (Actual); Status verified 2024-02

CONDITIONS: Brain Injuries; Brain Injuries, Traumatic; Brain Injuries, Vascular
Keywords: acquired brain injury; traumatic; virtual reality; cognitive function; rehabilitation; disability; lower limb; personalized medicine
MeSH Terms: conditions — Brain Injuries; Brain Injuries, Traumatic; Cerebrovascular Trauma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (no visual feedback-visual feedback) (Experimental): Participants in group A (6 patients with sABI and 6 healthy controls), will perform a single rehabilitation session with OMEGO®. In total, they will perform 18 minutes divided as follows: 5 minutes of treatment with OMEGO® without visual feedback, 3 minutes of break, and additional 5 minutes of treatment with OMEGO® plus visual feedback
  Interventions: Device: OMEGO®
- Group B (visual feedback-no visual feedback) (Experimental): Participants in group B (6 patients with sABI and 6 healthy controls), will perform a single rehabilitation session with OMEGO®. In total, they will perform 18 minutes divided as follows: 5 minutes of treatment with OMEGO® plus visual feedback, 3 minutes of break, and additional 5 minutes of treatment with OMEGO® without visual feedback
  Interventions: Device: OMEGO®

INTERVENTIONS:
Device: OMEGO® — Lower limb rehabilitation with and without visual feedback

SUMMARY:
Severe Acquired Brain Injury (sABI) is defined as "an encephalic impairment that occurs after birth and is not related to a congenital or degenerative disease.

This impairment may be temporary, or permanent, and cause partial or functional disability or psychosocial distress." In Italy there are at least 10-15 new cases of sABI per year per 100,000 inhabitants; the estimated prevalence is about 150,000 cases per year. Often, people with sABI present focal neurological deficits, including alterations in strength, sensitivity, coordination and gait.

Most of the rehabilitation protocols for people with sABI are derived from post-stroke studies, caused by lack of evidence on specific rehabilitation of people with sABI. Rehabilitation of people with sABI should begin as soon as possible, to prevent the onset of retractions and decubitus, and to regain joint mobility, strength, and coordination.

OMEGO® (Tyromotion) is a newly developed device used in lower extremity rehabilitation, that provides visual and auditory feedback.

Specifically, OMEGO® contains several games developed to enhance and promote learning behaviors, that simulate activities of daily living. The use of devices such as cycle ergometers is recommended in the rehabilitation of people with sABI; however, there are no studies demonstrating the effect of cycle ergometer training in association with visual feedback.

The purpose of this study is to evaluate, both in people without apparent pathology (hereafter identified as "healthy") and in people with sABI, whether visual feedback during OMEGO® exercise modifies brain connectivity, emotional drive, and lower limb performance during a lower limb-specific motor rehabilitation task.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis os severe Acquired Brain Injury (sABI)
* Trunk Control Test score greater or equal to 48
* Motricity Index Lower Limb score greater or equal to 18
* Clinical stability
* Patient/Caregiver ability to understand ans sing the informed consent

Exclusion Criteria:

* Disorder of consciousness (mininally concious state or vegetative state)
* severe visual impairment (central or peripheral, prior or acquired after the scute event)
* presence of severe cognitive impairment
* presence of global aphasia or presence of severe apraxia

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2020-10-13 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-10-31 (Actual)

PRIMARY OUTCOMES:
Change of Symmetry after the performance of the motor task | Change from baseline at T4 [after 18 minutes]
  The symmetry between lower limbs will be evaluated, comparing the percentage of movement between limbs.

SECONDARY OUTCOMES:
Brain connectivity | Baseline [T0]; after 5 minutes [training1, T1], after 8 minutes [rest, T2]; after 13 minutes [training2,T3] and after 18 minutes [rest, T4]
  Assessment of brain connectivity will be performed by evaluating the EEG
Electrodermal activity | Baseline [T0]; after 5 minutes [training1, T1], after 8 minutes [rest, T2]; after 13 minutes [training2,T3] and after 18 minutes [rest, T4]
  Electrodermal activity assessment will be performed using the E4 wearable medical device (Empatica)
Heart Rate Variability | Baseline [T0]; after 5 minutes [training1, T1], after 8 minutes [rest, T2]; after 13 minutes [training2,T3] and after 18 minutes [rest, T4]
  Heart Rate Variability assessment will be performed using the E4 wearable medical device (Empatica)
Change of Proprioception | Change from baseline at T4 [after 18 minutes]
  The proprioception of lower limbs will be evaluated by asking the patient to reach with the lower limb an indicated position

CONTACTS AND LOCATIONS:
Overall Officials: Augusto Fusco, MD, phD, Study Director — Fondazione Policlinico Universitaria A. Gemelli IRCCS
Locations (1):
- UOC Neuroriabilitazione ad Alta Intensità, Fondazione Policlinico Universitario A. Gemelli IRCCS, Rome, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Maegele M. Traumatic brain injury in 2017: exploring the secrets of concussion. Lancet Neurol. 2018 Jan;17(1):13-15. doi: 10.1016/S1474-4422(17)30419-2. Epub 2017 Dec 16. No abstract available. PMID 29262993
- [Background] Horn SD, Corrigan JD, Dijkers MP. Traumatic Brain Injury Rehabilitation Comparative Effectiveness Research: Introduction to the Traumatic Brain Injury-Practice Based Evidence Archives Supplement. Arch Phys Med Rehabil. 2015 Aug;96(8 Suppl):S173-7. doi: 10.1016/j.apmr.2015.03.027. PMID 26212395
- [Background] Aulisio MC, Han DY, Glueck AC. Virtual reality gaming as a neurorehabilitation tool for brain injuries in adults: A systematic review. Brain Inj. 2020 Aug 23;34(10):1322-1330. doi: 10.1080/02699052.2020.1802779. Epub 2020 Aug 13. PMID 32791020
- [Background] Nudo RJ. Adaptive plasticity in motor cortex: implications for rehabilitation after brain injury. J Rehabil Med. 2003 May;(41 Suppl):7-10. doi: 10.1080/16501960310010070. PMID 12817650
- [Background] Laudisio A, Giovannini S, Finamore P, Loreti C, Vannetti F, Coraci D, Incalzi RA, Zuccal G, Macchi C, Padua L; Mugello Study Working Group. Muscle strength is related to mental and physical quality of life in the oldest old. Arch Gerontol Geriatr. 2020 Jul-Aug;89:104109. doi: 10.1016/j.archger.2020.104109. Epub 2020 May 15. PMID 32460125
- [Background] Castelli L, De Giglio L, Haggiag S, Traini A, De Luca F, Ruggieri S, Prosperini L. Premorbid functional reserve modulates the effect of rehabilitation in multiple sclerosis. Neurol Sci. 2020 May;41(5):1251-1257. doi: 10.1007/s10072-019-04237-z. Epub 2020 Jan 9. PMID 31919697
- [Background] Levin MF, Weiss PL, Keshner EA. Emergence of virtual reality as a tool for upper limb rehabilitation: incorporation of motor control and motor learning principles. Phys Ther. 2015 Mar;95(3):415-25. doi: 10.2522/ptj.20130579. Epub 2014 Sep 11. PMID 25212522
- [Background] Mukamel R, Ekstrom AD, Kaplan J, Iacoboni M, Fried I. Single-neuron responses in humans during execution and observation of actions. Curr Biol. 2010 Apr 27;20(8):750-6. doi: 10.1016/j.cub.2010.02.045. Epub 2010 Apr 8. PMID 20381353
- [Background] Laver KE, Lange B, George S, Deutsch JE, Saposnik G, Crotty M. Virtual reality for stroke rehabilitation. Cochrane Database Syst Rev. 2017 Nov 20;11(11):CD008349. doi: 10.1002/14651858.CD008349.pub4. PMID 29156493
- [Background] Milgram, P.; Kishino, F. A taxonomy of mixed reality visual displays. IEICE Trans. Inform. Syst. 1994, 77, 1321-1329.
- [Background] Yin C, Hsueh YH, Yeh CY, Lo HC, Lan YT. A Virtual Reality-Cycling Training System for Lower Limb Balance Improvement. Biomed Res Int. 2016;2016:9276508. doi: 10.1155/2016/9276508. Epub 2016 Mar 6. PMID 27034953
- [Background] Kleim JA, Jones TA. Principles of experience-dependent neural plasticity: implications for rehabilitation after brain damage. J Speech Lang Hear Res. 2008 Feb;51(1):S225-39. doi: 10.1044/1092-4388(2008/018). PMID 18230848
- [Background] Padua L, Imbimbo I, Aprile I, Loreti C, Germanotta M, Coraci D, Piccinini G, Pazzaglia C, Santilli C, Cruciani A, Carrozza MC; FDG Robotic Rehabilitation Groupdagger. Cognitive reserve as a useful variable to address robotic or conventional upper limb rehabilitation treatment after stroke: a multicentre study of the Fondazione Don Carlo Gnocchi. Eur J Neurol. 2020 Feb;27(2):392-398. doi: 10.1111/ene.14090. Epub 2019 Oct 18. PMID 31536677
- [Background] Banz R, Bolliger M, Colombo G, Dietz V, Lunenburger L. Computerized visual feedback: an adjunct to robotic-assisted gait training. Phys Ther. 2008 Oct;88(10):1135-45. doi: 10.2522/ptj.20070203. Epub 2008 Sep 4. PMID 18772279